CLINICAL TRIAL: NCT03308370
Title: Evaluation of the Therapeutic Effect of Platelet Rich Plasma in Melasma
Brief Title: Platelet Rich Plasma in Treatment of Melasma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, A Ghazally, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETEPRPM
Record Dates: First submitted 2017-10-07; First posted 2017-10-12 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Melasma; Platelet Rich Plasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Platelet rich plasma (Experimental): intradermal injection of 5 ml of autologous platelet rich plasma in the lesional skin of the face of 20 melasma patients every 4 weeks for 3 times
  Interventions: Biological: Platelet rich plasma

INTERVENTIONS:
Biological: Platelet rich plasma — 10 ml of blood will be drawn from the patients on an anticoagulant then it will be centrifuged to get platelet rich plasma that will be injected in the melasma lesions of the patients after its activation with calcium chloride.

SUMMARY:
Melasma is a common acquired disorder characterized by symmetric, hyperpigmented patches with an irregular outline, occurring most commonly on the face. The therapy for melasma has always been challenging and discouraging. Platelet rich plasma has been used over the last several years as an effective treatment in various surgical and medical ﬁelds. In recent years, Platelet rich plasma has also started to be used in the field of cosmetology. This study is designed to evaluate the therapeutic effect of platelet rich plasma in melasma.

DETAILED DESCRIPTION:
Melasma is a pigmentary disorder that can be disfiguring and can cause to significant emotional stresses for sufferers, for which a universally effective treatment is still lacking. Platelet rich plasma is commonly used in dermatology and plastic surgery, especially for treating chronic wounds, ulcers, and burns. The most important contents of platelets are contained in the α-granules. Some of the bioactive substances present in the α-granules include platelet-derived growth factor, transforming growth factor -β1 and -β2epidermal growth factor, and mitogenic growth factors such as platelet-derived angiogenesis factor and fibrinogen.

transforming growth factor -β1 decreases melanogenesis via delayed extracellular signal-regulated kinase activation. The regression of melasma in a 27-years-old woman after injecting platelet rich plasma for skin rejuvenation was observed, but controlled clinical trials are still lacking to confirm this preliminary observation.

ELIGIBILITY:
Inclusion Criteria:

* patients with melasma 18 years old or more

Exclusion Criteria:

* Patients less than 18 years.
* Pregnant females and females on oral contraceptive pills.
* Patients with a history of hypertrophic scars or keloids.
* Patients with recurrent herpes infection or with present cutaneous infection and those with facial cancer.
* Patients with blood disorders and platelet abnormalities and chronic liver disease.
* Patients using systemic chemotherapy, anticoagulation therapy and antiplatelet agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-07 (Estimated)

PRIMARY OUTCOMES:
clinical improvement of melasma | 3 months
  evaluation of the degree of clinical improvement of melasma by using platelet rich plasma

SECONDARY OUTCOMES:
evaluation of transforming growth factor beta expression in the melasma skin | 3 months
  compare the intensity of immunohistochemical expression of transforming growth factor beta in skin biopsies taken from the the lesional melasma skin ( of participants who accept only) before and after treatment with platelet rich plasma The results will be scored as follows: 0 for negative staining, 1+ for weak staining, 2+ for moderate staining intensity, and 3+ for strong positive staining.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa H Ghazally, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut university hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Grimes PE. Melasma. Etiologic and therapeutic considerations. Arch Dermatol. 1995 Dec;131(12):1453-7. doi: 10.1001/archderm.131.12.1453. PMID 7492140
- [Background] Cayirli M, Caliskan E, Acikgoz G, Erbil AH, Erturk G. Regression of melasma with platelet-rich plasma treatment. Ann Dermatol. 2014 Jun;26(3):401-2. doi: 10.5021/ad.2014.26.3.401. Epub 2014 Jun 12. No abstract available. PMID 24966645
- [Background] Kim DS, Park SH, Park KC. Transforming growth factor-beta1 decreases melanin synthesis via delayed extracellular signal-regulated kinase activation. Int J Biochem Cell Biol. 2004 Aug;36(8):1482-91. doi: 10.1016/j.biocel.2003.10.023. PMID 15147727